CLINICAL TRIAL: NCT00690521
Title: A Comparison of Hydrochlorothiazide and Metolazone in Combination With Furosemide in Congestive Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Joe R. Anderson, Principal Investigator, University of New Mexico
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HRRC 03-477
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Congestive Heart Failure
Keywords: congestive heart failure; diuretics; combination
MeSH Terms: conditions — Heart Failure | interventions — Hydrochlorothiazide; Metolazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Furosemide and hydrochlorothiazide (Experimental): A randomized, double-blind, crossover study designed to compare the efficacy of hydrochlorothiazide in combination with stable doses of furosemide in congestive heart failure patients.
  Interventions: Drug: Treatment of Furosemide + Hydrochlorothiazide
- Furosemide and metolazone (Experimental): A randomized, double-blind, crossover study designed to compare the efficacy of metolazone in combination with stable doses of furosemide in congestive heart failure patients.
  Interventions: Drug: Treatment of Furosemide + Metolazone

INTERVENTIONS:
Drug: Treatment of Furosemide + Hydrochlorothiazide — A randomized, double-blind, crossover study designed to compare the efficacy of hydrochlorothiazide in combination with stable doses of furosemide in congestive heart failure patients.
  Arms: Furosemide and hydrochlorothiazide
Drug: Treatment of Furosemide + Metolazone — A randomized, double-blind, crossover study designed to compare the efficacy of metolazone in combination with stable doses of furosemide in congestive heart failure patients.
  Arms: Furosemide and metolazone

SUMMARY:
Objective: To establish which combination of diuretics is the most effective in promoting diuresis in congestive heart failure patients. Secondary Objectives: To determine the duration of action of furosemide as monotherapy and in combination hydrochlorothiazide with metolazone. To determine the effect of diuretic combination therapy on neurohormonal activation. Background: Diuretic resistance occurs when a potent diuretic drug, such as furosemide, is given in therapeutic doses and fails to reduce extracellular fluid volume to the desired level in an edematous patient. Studies have shown that metolazone and hydrochlorothiazide have demonstrated a synergistic response when used in combination with furosemide in congestive heart failure patients. The current guidelines for treating diuretic resistance in congestive heart failure patients recommend the metolazone-furosemide combination. However, there is no evidence to conclude that this combination is superior to hydrochlorothiazide-furosemide in increasing diuresis. Methods: Study to compare the efficacy of hydrochlorothiazide with metolazone in combination with stable doses of furosemide in 13 patients with congestive heart failure. The primary endpoint will be change in urinary output. Secondary endpoints will be changes in weight, neurohormones (angiotensin II, catecholamines, brain natriuretic peptide, aldosterone), and electrocardiographic parameters of ventricular instability. Study procedures will be performed at the UNM General Clinical Research Center. Patients will be hospitalized for 2 separate 4-day admissions, separated by a 1-week washout period. At each admission each patient will receive furosemide in combination with either metolazone or hydrochlorothiazide (metolazone for one admission and hydrochlorothiazide for the other). Following administration of combination therapy, blood and urine samples will be collected throughout the day to chart the onset and magnitude of effect of each treatment regimen. Various hemodynamic, renal, endocrine, and neurohormonal parameters will be assesed as will the effect of each combination treatment on ventricular instability using 12-lead electrocardiography. Data will be analyzed using ANOVA to compare changes from baseline and the Student t-test to analyze intertreatment differences.

All statistical analysis will be performed using SAS v6.12.d

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Diagnosis of chronic congestive heart failure with an ejection fraction ≤45%
* Currently on a stable regimen of furosemide consisting of a daily dose of at least 80 mg for at least two weeks.
* Patients receiving ACE-inhibitors and/or beta-blockers must be taking these medications for at least two weeks in stable doses.

Exclusion Criteria:

* Renal dysfunction (serum creatinine >2 mg/dl or creatinine clearance of <30 ml/min as calculated by the Cockroft and Gault equation)
* Hepatic dysfunction (AST and ALT >3 times the upper limit of the normal)
* Hypokalemia (<4.0 mg/dl)
* Concomitant treatment with any diuretic other than furosemide (with the exception of spironolactone).

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-10-26 (Actual); Primary Completion 2009-11-10 (Actual); Study Completion 2009-11-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Of New Mexico Hospital, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8 patients enrolled and received drug treatment.
Groups:
- Arm 1-Furosemide + Hydrochlorothiazide Then Furosemide + Metolazone: A Randomized, double-blind, crossover study designed to compare the efficacy of furosemide in combination with hydrochlorothiazide or metolazone in congestive heart failure patients.
  First Intervention- Furosemide and Hydrochlorothiazide (4 days) Washout (7 days) Second Intervention-Furosemide + Metolazone (4 days)
  Combined results for both therapies are being reported since it cannot be determined which arm/group was assigned to Hydrochlorothiazide or metolazone
- Arm-2 Furosemide + Metolazone Then Furosemide + Hydrochlorothiazide: A Randomized, double-blind, crossover study designed to compare the efficacy of furosemide in combination with hydrochlorothiazide or metolazone in congestive heart failure patients.
  First Intervention-Furosemide + Metolazone (4 days) Washout (7 days) Second Intervention-Furosemide and Hydrochlorothiazide (4 days)
  Combined results for both therapies are being reported since it cannot be determined which arm/group was assigned to Hydrochlorothiazide or metolazone
Period: First Intervention (4 Days)
Arm/Group | Arm 1-Furosemide + Hydrochlorothiazide Then Furosemide + Metolazone | Arm-2 Furosemide + Metolazone Then Furosemide + Hydrochlorothiazide
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: Washout (7 Days)
Arm/Group | Arm 1-Furosemide + Hydrochlorothiazide Then Furosemide + Metolazone | Arm-2 Furosemide + Metolazone Then Furosemide + Hydrochlorothiazide
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: Second Intervention (4 Days)
Arm/Group | Arm 1-Furosemide + Hydrochlorothiazide Then Furosemide + Metolazone | Arm-2 Furosemide + Metolazone Then Furosemide + Hydrochlorothiazide
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Drug A followed by Drug B.
Groups:
- Arm 1: A Randomized, double-blind, crossover study designed to compare the efficacy of furosemide in combination with hydrochlorothiazide or metolazone in congestive heart failure patients.
  First Intervention with Furosemide and Hydrochlorothiazide (4 days), Washout (7 days), and Second Intervention with Furosemide + Metolazone(4 days).
Arm/Group | Arm 1
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 3
  Other | 5

OUTCOME MEASURES:

1. Primary Outcome: Participants With Change in Urinary Output
Time Frame: First Intervention (4 days), Washout (7 days), and Second Intervention (4 days)
Measure: Number; unit: participants
Groups:
- Arm1- Furosemide and Hydrochlorothiazide Then Furosemide + Metolazone: A Randomized, double-blind, crossover study designed to compare the efficacy of furosemide in combination with hydrochlorothiazide or metolazone in congestive heart failure patients.
  First Intervention-Furosemide and Hydrochlorothiazide (4 days) Washout (7 days) Second Intervention-Furosemide + Metolazone (4 days)
  Combined results for both therapies are being reported since it cannot be determined which arm/group was assigned to Hydrochlorothiazide or metolazone
- Arm2-Furosemide and Metolazone Then Furosemide and Hydrochlorothiazide: A Randomized, double-blind, crossover study designed to compare the efficacy of furosemide in combination with hydrochlorothiazide or metolazone in congestive heart failure patients.
  First Intervention-Furosemide and Metolazone (4 days) Washout (7 days) Second Intervention-Furosemide and Hydrochlorothiazide (4 days),
  Combined results for both therapies are being reported since it cannot be determined which arm/group was assigned to Hydrochlorothiazide or metolazone
Arm/Group | Arm1- Furosemide and Hydrochlorothiazide Then Furosemide + Metolazone | Arm2-Furosemide and Metolazone Then Furosemide and Hydrochlorothiazide
Number analyzed (Participants) | 4 | 4
participants
  First Intervention (4 days) | 4 | 4
  Washout (7 days) | 4 | 4
  Second Intervention (4 days) | 4 | 4

ADVERSE EVENTS:
Groups:
- Arm 1-First Intervention-Furosemide + Hydrochlorothiazide; Arm 1-Second Intervention-Furosemide + Metolazone: A Randomized, double-blind, crossover study designed to compare the efficacy of furosemide in combination with hydrochlorothiazide or metolazone in congestive heart failure patients.
  First Intervention-Furosemide and Hydrochlorothiazide (4 days) Washout (7 days) Second Intervention with Furosemide + Metolazone (4 days)
  Combined results for both therapies are being reported since it cannot be determined which arm/group was assigned to Hydrochlorothiazide or metolazone.
- Arm 2-First Intervention-Furosemide + Metolazone; Arm 2-Second Intervention-Furosemide + Hydrochlorothiazide: A Randomized, double-blind, crossover study designed to compare the efficacy of furosemide in combination with hydrochlorothiazide or metolazone in congestive heart failure patients.
  First Intervention- Furosemide + Metolazone (4 days) Washout (7 days) Second Intervention with Furosemide + Hydrochlorothiazide (4 days)
  Combined results for both therapies are being reported since it cannot be determined which arm/group was assigned to Hydrochlorothiazide or metolazone.
Arm/Group | Arm 1-First Intervention-Furosemide + Hydrochlorothiazide | Arm 1-Second Intervention-Furosemide + Metolazone | Arm 2-First Intervention-Furosemide + Metolazone | Arm 2-Second Intervention-Furosemide + Hydrochlorothiazide
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2007-05-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT00690521/Prot_000.pdf
  • Informed Consent Form (2009-06-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT00690521/ICF_001.pdf